CLINICAL TRIAL: NCT05282121
Title: Randomised, Open-label and Parallel Group Trial to Investigate the Effects of Oral BI 685509 Alone or in Combination With Empagliflozin on Portal Hypertension After 8 Weeks Treatment in Patients With Clinically Significant Portal Hypertension (CSPH) in Compensated Cirrhosis
Brief Title: A Study to Test Whether BI 685509 Alone or in Combination With Empagliflozin Helps People With Liver Cirrhosis Caused by Viral Hepatitis or Non-alcoholic Steatohepatitis (NASH) Who Have High Blood Pressure in the Portal Vein (Main Vessel Going to the Liver)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1366-0029; 2021-005171-40 (EudraCT Number); 2023-504257-12-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2022-03-14; First posted 2022-03-16 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Liver Diseases; Hypertension, Portal
MeSH Terms: conditions — Liver Diseases; Hypertension, Portal | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Patients with HBV - avenciguat (Experimental): Patients with Hepatitis B Virus (HBV) were administered one film-coated tablet of avenciguat orally twice a day. The two doses were ideally taken at least 10 hours apart. The starting dose was 1 milligram (mg), which, if tolerated, was up-titrated to 2 mg one week later. If this dose was also tolerated, a second up-titration to 3 mg occured after another week. Patients remained on the highest dose for the remainder of the treatment period, until 8 weeks of treatment.
  Interventions: Drug: Avenciguat
- Patients with HCV - avenciguat (Experimental): Patients with Hepatitis C Virus (HCV) were administered one film-coated tablet of avenciguat orally twice a day. The two doses were ideally taken at least 10 hours apart. The starting dose was 1 milligram (mg), which, if tolerated, was up-titrated to 2 mg one week later. If this dose was also tolerated, a second up-titration to 3 mg occured after another week. Patients remained on the highest dose for the remainder of the treatment period, until 8 weeks of treatment.
  Interventions: Drug: Avenciguat
- Patients with NASH with or without T2DM - avenciguat (Experimental): Patients with Non-Alcoholic Steatohepatitis (NASH) with or without type 2 Diabetes Mellitus (T2DM) were administered one film-coated tablet of avenciguat orally twice a day. The two doses were ideally taken at least 10 hours apart. The starting dose was 1 milligram (mg), which, if tolerated, was up-titrated to 2 mg one week later. If this dose was also tolerated, a second up-titration to 3 mg occured after another week. Patients remained on the highest dose for the remainder of the treatment period, until 8 weeks of treatment.
  Interventions: Drug: Avenciguat
- Patients with NASH with T2DM - avenciguat + empagliflozin (Experimental): Patients with Non-Alcoholic Steatohepatitis (NASH) with type 2 Diabetes Mellitus (T2DM) were administered one film-coated tablet of avenciguat orally twice a day. The two doses were ideally taken at least 10 hours apart. The starting dose was 1 milligram (mg), which, if tolerated, was up-titrated to 2 mg one week later. If this dose was also tolerated, a second up-titration to 3 mg occured after another week. Patients remained on the highest dose for the remainder of the treatment period, until 8 weeks of treatment.
  Patients were additionally administered one 10 mg film-coated tablet of empagliflozin orally once a day.
  Interventions: Drug: Avenciguat; Drug: Empagliflozin

INTERVENTIONS:
Drug: Avenciguat — one film-coated tablet orally twice a day, at least 10 hours apart. The starting dose (1 mg) was up-titrated up to 3 mg
  Other Names: BI 685509
Drug: Empagliflozin — one 10 mg film-coated tablet of orally once a day
  Arms: Patients with NASH with T2DM - avenciguat + empagliflozin

SUMMARY:
This study is open to adults with liver cirrhosis caused by hepatitis B, hepatitis C or nonalcoholic steatohepatitis (NASH). People can join this study if they have high blood pressure in the portal vein (main vessel going to the liver).

The purpose of this study is to find out whether a medicine called Avenciguat (BI 685509) taken alone or in combination with a medicine called empagliflozin helps people with this condition.

Participants take Avenciguat (BI 685509) as tablets twice a day for 8 weeks. Half of the participants with NASH who also have type 2 diabetes take empagliflozin as tablets once a day in addition to Avenciguat (BI 685509).

Participants are in the study for about 3 months. During this time, they visit the study site about 10 times. At 2 of the visits, the doctors check the pressure in a liver vein to see whether the treatment works. This is done with a catheter (a long thin tube) and gives information about the pressure in the portal vein. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Male or female who is ≥ 18 (or who is of legal age in countries where that is greater than 18) and ≤ 75 years old at screening (Visit 1a)
* Clinical signs of Clinically Significant Portal Hypertension (CSPH) as described by either one of the points below. Each trial patient must have a gastroscopy during the screening period (Visit 1b) or within 6 months prior to screening (Visit 1b).

  * documented endoscopic proof of oesophageal varices and / or gastric varices at screening (Visit 1b) or within 6 months prior to screening (Visit 1b)
  * documented endoscopic-treated oesophageal varices as preventative treatment
* CSPH defined as baseline Hepatic Venous Pressure Gradient (HVPG) ≥ 10 mmHg (measured at Visit 1c), based on a local interpretation of the pressure tracing
* Diagnosis of compensated cirrhosis due to Hepatitis C virus (HCV), Hepatitis B virus (HBV), or Non-Alcoholic Steatohepatitis (NASH) with or without Type 2 Diabetes Melitus (T2DM). Diagnosis of cirrhosis must be based on histology (historical data is acceptable) or on clinical evidence of cirrhosis (e.g. platelet count < 150 x 109/L [150 x 103/microlitre (μL)], nodular liver surface on imaging or splenomegaly etc.) Diagnosis of NASH based on either i. Current or historic histological diagnosis of NASH OR steatosis OR ii. Clinical diagnosis of NASH based on historic or current imaging diagnosis of fatty liver (Fibroscan, Ultrasound (US), Magnetic Resonance Imaging (MRI), Computed Tomography (CT)) AND at least 2 current or historic comorbidities of the metabolic syndrome (overweight/obesity, T2DM, hypertension, hyperlipidemia)
* Willing and able to undergo HVPG measurements per protocol (based on Investigator judgement)
* If receiving statins must be on a stable dose for at least 3 months prior to screening (Visit 1b), with no planned dose change throughout the trial
* If receiving treatment with Non-Selective Beta-Blocker (NSBBs) or carvedilol must be on a stable dose for at least 1 months prior to screening (Visit 1b), with no planned dose change throughout the trial
* Further inclusion criteria apply

Exclusion Criteria:

* Previous clinically significant decompensation events (e.g. ascites [more than perihepatic ascites], Variceal Haemorrhage (VH) and / or overt / apparent Hepatic Encephalopathy (HE))
* History of other forms of chronic liver disease (e.g. alcohol-related liver disease (ARLD), autoimmune liver disease, primary biliary sclerosis, primary sclerosing cholangitis, Wilson's disease, haemachromatosis, alpha-1 antitrypsin [A1At] deficiency)
* Patients without adequate treatment for HBV, HCV or NASH as per local guidance (e.g. antiviral therapy for chronic HBV or HCV infection or lifestyle modification in NASH)

  * if received curative anti-viral therapy for HCV, no sustained virological response (SVR) or SVR sustained for less than 2 years prior to screening or if HCV Ribonucleic Acid (RNA) detectable
  * If receiving anti-viral therapy for HBV, less than 6 months on a stable dose prior to screening, with planned dose change during the trial or HBV deoxyribonucleic acid (DNA) detectable
  * Weight change ≥ 5% within 6 months prior screening
* Must take, or wishes to continue the intake of, restricted concomitant therapy or any concomitant therapy considered likely (based on Investigator judgement) to interfere with the safe conduct of the trial
* Systolic Blood Pressure (SBP) < 100 mmHg and Diastolic Blood Pressure (DBP) < 70 mmHg at screening (Visit 1a)
* Model of End-stage Liver Disease (MELD) score of > 15 at screening (Visit 1a), calculated by the central laboratory
* Hepatic impairment defined as a Child-Turcotte-Pugh score ≥ B8 at screening (Visit 1a), calculated by the site, using central laboratory results
* Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 5 times upper limit of normal (ULN) at screening (Visit 1a), measured by the central laboratory
* Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (4):
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Floridian Clinical Research-Miami Lakes-68368, Miami Lakes, Florida
  - American Research Corporation, San Antonio, Texas
- Argentina (2):
  - Hospital Britanico de Buenos Aires, CABA
  - Hospital Italiano de Buenos Aires, CABA
- AKH - Medical University of Vienna, Vienna, Austria
- Edegem - UNIV UZ Antwerpen, Edegem, Belgium
- Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec, Canada
- China (4):
  - Beijing Friendship Hospital, Beijing
  - NanFang Hosptial, Guangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
- Hvidovre Hospital, Hvidovre, Denmark
- France (2):
  - HOP Beaujon, Clichy
  - HOP Rangueil, Toulouse
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Münster, Münster
- Israel (2):
  - Rambam Medical Center, Haifa
  - Western Galilee Hospital, Nahariya
- Italy (3):
  - Ospedale Civile di Baggiovara, Baggiovara (MO)
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - Policlinico "Paolo Giaccone", Palermo
- Japan (2):
  - National Hospital Organization Yokohama Medical Center, Kanagawa, Yokohama
  - Osaka Metropolitan University Hospital, Osaka, Osaka
- Amsterdam UMC, location VUMC, Amsterdam, Netherlands
- Regional Institute of Gastroenterology Hepatology "Prof. Dr. O. Fodor", Cluj-Napoca, Romania
- Singapore General Hospital, Singapore, Singapore
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Reiberger T, Berzigotti A, Trebicka J, Ertle J, Gashaw I, Swallow R, Tomisser A. The rationale and study design of two phase II trials examining the effects of BI 685,509, a soluble guanylyl cyclase activator, on clinically significant portal hypertension in patients with compensated cirrhosis. Trials. 2023 Apr 24;24(1):293. doi: 10.1186/s13063-023-07291-3. PMID 37095557
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomised, open-label, parallel-group multinational phase II trial was conducted to investigate the effects of oral avenciguat (BI 685509) alone and in combination with empagliflozin on portal hypertension after 8 weeks treatment in patients with clinically significant portal hypertension (CSPH) in compensated cirrhosis.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any entry criteria were violated.
Period: Overall Study
Arm/Group | Patients With HBV - Avenciguat | Patients With HCV - Avenciguat | Patients With NASH With or Without T2DM - Avenciguat | Patients With NASH With T2DM - Avenciguat + Empagliflozin
Started | 14 | 13 | 38 | 25
Completed | 12 | 10 | 30 | 22
Not Completed | 2 | 3 | 8 | 3
Not completed — Adverse Event | 1 | 1 | 4 | 1
Not completed — Study Terminated by Sponsor | 1 | 2 | 2 | 2
Not completed — Other than listed | 0 | 0 | 1 | 0
Not completed — No reason available | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all patients who were enrolled or randomised to the trial medication and were treated with at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With HBV - Avenciguat | Patients With HCV - Avenciguat | Patients With NASH With or Without T2DM - Avenciguat | Patients With NASH With T2DM - Avenciguat + Empagliflozin | Total
Number analyzed (Participants) | 14 | 13 | 38 | 25 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (12.0) | 60.3 (7.2) | 62.6 (7.5) | 64.1 (5.6) | 60.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 23 | 16 | 45
  Male | 14 | 7 | 15 | 9 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 14 | 14 | 34
  Not Hispanic or Latino | 12 | 9 | 24 | 11 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 9 | 0 | 2 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 4 | 13 | 35 | 23 | 75
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Hepatic Venous Pressure Gradient (HVPG) [Mean (Standard Deviation); unit: millimetre of mercury (mmHg)] — HVPG measurement at baseline was performed before the first intake of trial medication. Population: Treated set. Only patients with available HVPG measurements were included.
  millimetre of mercury (mmHg)
    number analyzed (Participants) | 14 | 13 | 37 | 24 | 88
    (all) | 13.68 (3.94) | 12.10 (2.51) | 15.46 (4.53) | 15.28 (3.70) | 14.63 (4.10)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in HVPG From Baseline (Measured in mmHg) After 8 Weeks of Treatment
Description: Percentage change in Hepatic Venous Pressure Gradient (HVPG) from baseline (measured in millimetre of mercury [mmHg]) after 8 weeks of treatment is reported. Adjusted mean (Least Square Mean) was calculated using an analysis of covariance (ANCOVA) model without imputing the missing data. The model included treatment as fixed classification effects, and baseline HVPG as a linear covariate. The random error was assumed to be normally distributed with mean 0 and variance σ².
Time Frame: Before the first intake of trial medication (baseline), and after 8 weeks of treatment.
Population: Full analysis set (FAS): this analysis set includes all enrolled or randomised patients who received at least one dose of trial medication and have a baseline measurement for the primary endpoint recorded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of change in HVPG
Arm/Group | Patients With HBV - Avenciguat | Patients With HCV - Avenciguat | Patients With NASH With or Without T2DM - Avenciguat | Patients With NASH With T2DM - Avenciguat + Empagliflozin
Number analyzed (Participants) | 14 | 13 | 37 | 24
Percentage of change in HVPG | -16.06 (6.66) | -5.81 (7.09) | 3.83 (4.25) | 3.27 (5.08)

2. Secondary Outcome: Occurrence of a Response, Which is Defined as > 10% Reduction From Baseline HVPG (Measured in mmHg) After 8 Weeks of Treatment
Description: Occurrence of a response, which is defined as > 10% reduction from baseline HVPG (measured in mmHg) after 8 weeks of treatment is reported.
Time Frame: Before the first intake of trial medication (baseline), and after 8 weeks of treatment.
Population: Full analysis set (FAS): this analysis set includes all enrolled or randomised patients who received at least one dose of trial medication and have a baseline measurement for the primary endpoint recorded. Only patients with a HVPG measurement at week 8 are reported.
Measure: Number; unit: Count of participants
Arm/Group | Patients With HBV - Avenciguat | Patients With HCV - Avenciguat | Patients With NASH With or Without T2DM - Avenciguat | Patients With NASH With T2DM - Avenciguat + Empagliflozin
Number analyzed (Participants) | 11 | 10 | 27 | 19
Count of participants | 9 | 2 | 9 | 4

3. Secondary Outcome: Occurrence of One or More Decompensation Events (i.e. Ascites, VH, and / or Overt HE) During the 8-week Treatment Period
Description: Occurrence of one or more decompensation events (i.e. ascites, Variceal Haemorrhage [VH], and / or overt Hepatic Encephalopathy [HE]) during the 8-week treatment period is reported.
Time Frame: From first intake of study medication, until last intake of study medication plus 7 days, up to approximately 10 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Count of participants
Arm/Group | Patients With HBV - Avenciguat | Patients With HCV - Avenciguat | Patients With NASH With or Without T2DM - Avenciguat | Patients With NASH With T2DM - Avenciguat + Empagliflozin
Number analyzed (Participants) | 14 | 13 | 38 | 25
Count of participants | 1 | 0 | 4 | 1

4. Secondary Outcome: Occurrence of CTCAE Grade 3 (or Higher) Hypotension or Syncope Based on Investigator Judgement, During the 8-week Treatment Period
Description: Occurrence of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 (or higher) hypotension or syncope based on Investigator judgement, during the 8-week treatment period is reported.
  The CTCAE grades are: 1 (mild Adverse Event [AE]), 2 (moderate AE), 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: From first intake of study medication, until last intake of study medication plus 7 days, up to approximately 10 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Count of participants
Arm/Group | Patients With HBV - Avenciguat | Patients With HCV - Avenciguat | Patients With NASH With or Without T2DM - Avenciguat | Patients With NASH With T2DM - Avenciguat + Empagliflozin
Number analyzed (Participants) | 14 | 13 | 38 | 25
Count of participants | 0 | 0 | 0 | 1

5. Secondary Outcome: Occurrence of Discontinuation Due to Hypotension or Syncope During the 8-week Treatment Period
Description: Occurrence of discontinuation of treatment with avenciguat due to hypotension or syncope during the 8-week treatment period is reported.
Time Frame: From first intake of study medication, until last intake of study medication plus 7 days, up to approximately 10 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Count of participants
Arm/Group | Patients With HBV - Avenciguat | Patients With HCV - Avenciguat | Patients With NASH With or Without T2DM - Avenciguat | Patients With NASH With T2DM - Avenciguat + Empagliflozin
Number analyzed (Participants) | 14 | 13 | 38 | 25
Count of participants | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first intake of study medication, until last intake of study medication plus 7 days, up to approximately 10 weeks (adverse events), or until end of study, up to 12 weeks (all-cause mortality).
Description: Treated set (TS): all patients who were enrolled or randomised to the trial medication and were treated with at least one dose of trial medication.
Arm/Group | Patients With HBV - Avenciguat | Patients With HCV - Avenciguat | Patients With NASH With or Without T2DM - Avenciguat | Patients With NASH With T2DM - Avenciguat + Empagliflozin
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/38 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/14 | 2/13 | 6/38 | 0/25
Other Adverse Events (participants affected / at risk) | 12/14 | 5/13 | 16/38 | 13/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With HBV - Avenciguat (N=14) | Patients With HCV - Avenciguat (N=13) | Patients With NASH With or Without T2DM - Avenciguat (N=38) | Patients With NASH With T2DM - Avenciguat + Empagliflozin (N=25)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With HBV - Avenciguat (N=14) | Patients With HCV - Avenciguat (N=13) | Patients With NASH With or Without T2DM - Avenciguat (N=38) | Patients With NASH With T2DM - Avenciguat + Empagliflozin (N=25)
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Temperature regulation disorder (General disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Electrocardiogram PR shortened (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 1 | 1 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT05282121/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT05282121/SAP_001.pdf